### **Statistical Analysis Plan**

Clinical trial protocol title: A Phase 1, Single-Blind, Randomized, Placebo

Controlled, Parallel-Group, Multiple-Dose Escalation

Study to Investigate Safety, Tolerability, and

Pharmacokinetics of Emodepside (BAY 44-4400) After

Oral Dosing in Healthy Male Subjects

HMR code: 16-021

Sponsor code: DNDI-EMO-02

EudraCT no: 2017-003020-75

CRO details: Hammersmith Medicines Research

Cumberland Avenue London NW10 7EW

Sponsor details: DNDi, Chemin Louis Dunant, 15,

1202 Geneva, Switzerland Phone: +41 22 906 9230

Issued: 29 August 2018

Version: 1

Based on: Protocol version 5, 25 July 2018

Number of pages: 70

Prepared by: Helen Topping

# **Table of contents**

| 1 | LIST | OF ABBREVIATIONS | 5 |
|----|------|-------------------------------------------------------|----|
| 2 | SIGN | NATURES | 7 |
| 3 | INTE | RODUCTION | 8 |
| 4 | STU | DY OBJECTIVE(S) AND ENDPOINT(S) | 8 |
| | 4.1 | Study Objective(s) | 8 |
| | | 4.1.1 Primary Objective(s) | 8 |
| | | 4.1.2 Secondary Objective(s) | 8 |
| | 4.2 | Study Endpoint(s) | 9 |
| | | 4.2.1 Primary Endpoint(s) | |
| | | 4.2.2 Secondary Endpoint(s) | |
| | 4.3 | Statistical Hypotheses | 10 |
| 5 | STU | DY DESIGN | 10 |
| 6 | TIM | E AND EVENTS TABLE | 12 |
| 7 | PLA] | NNED ANALYSES | 16 |
| | 7.1 | Interim Analyses | 16 |
| | | 7.1.1 Persons responsible for analysis | 16 |
| | 7.2 | Final Analysis | 16 |
| | | 7.2.1 Persons responsible for analysis | |
| 8 | SAM | PLE SIZE CONSIDERATIONS | 17 |
| | 8.1 | Sample Size Assumptions | 17 |
| 9 | ANA | LYSIS POPULATIONS | 17 |
| | 9.1 | Analysis Datasets | 17 |
| 10 | TRE | ATMENT COMPARISONS | 17 |
| 11 | GEN | ERAL CONSIDERATIONS FOR DATA ANALYSES | 17 |
| | 11.1 | Data Display Treatment and Other Subgroup Descriptors | 17 |
| | 11.2 | Conventions for Summary Statistics and Data Displays | 18 |
| 12 | DAT | A HANDLING CONVENTIONS | 18 |
| | 12.1 | Premature Withdrawal and Missing Data | 18 |
| | 12.2 | Derived and Transformed Data | 19 |
| | 12.3 | Assessment Windows | 19 |
| | 12.4 | Values of Potential Clinical Importance | 20 |
| 13 | STUI | DY POPULATION | 20 |
| | 13.1 | Disposition of Subjects | 20 |
| | 13.2 | Protocol Deviations | 21 |

| | 13.3 | Demographic and Baseline Characteristics | 21 |
|---|---|---|---|
| | 13.4 | Treatment Compliance | 21 |
| 14 | SAFE | ETY ANALYSES | 21 |
| | 14.1 | Extent of Exposure | 21 |
| | 14.2 | Adverse Events | 22 |
| | 14.3 | Deaths, Serious Adverse Events and Other Significant Adverse E | vents 22 |
| | 14.4 | Adverse Events Leading to Withdrawal from the Study | 22 |
| | 14.5 | Clinical Laboratory Evaluations | 23 |
| | 14.6 | Other Safety Measures | 23 |
| | | 14.6.1 Vital signs | 23 |
| | | 14.6.2 ECG | 23 |
| | | 14.6.3 Physical examination | 23 |
| | | 14.6.4 Neurological examination | 23 |
| | | 14.6.5 Ophthalmology examination | 24 |
| 15 | PHAR | RMACOKINETIC ANALYSES | 24 |
| | 15.1 | Plasma PK | 24 |
| | | 15.1.1 Pharmacokinetic Concentration Data | 24 |
| | | 15.1.2 Pharmacokinetic Parameters | 25 |
| | 15.2 | Urinary PK | 25 |
| 16 | PHAR | RMACODYNAMIC ANALYSES | 25 |
| 17 | REFE | ERENCES | 26 |
| 18 | ATTA | ACHMENTS | 26 |
| | 18.1 | Table of Contents for Data Display Specifications | 26 |
| | 18.2 | Data Display Specifications | 31 |
| | | 18.2.1 Table Outlines | 31 |
| | | 18.2.2 Figure Outlines | 42 |
| | | 18.2.3 Listing Outlines | 46 |
| APPI | ENDIX | A: LABORATORY RANGES | 58 |
| APPI | ENDIX | B: PHARMACOKINETIC ANALYSIS | 60 |
| 1 | CALC | CULATION METHODS | 60 |
| | 1.1 | Data Handling Conventions | 60 |
| | | 1.1.1 Actual v Planned Times | 60 |
| | | 1.1.2 Missing and BQL Concentrations | 60 |
| | 1.2 | AUC Calculations | 60 |
| | 1.3 | Lambda-z Calculations | 61 |
| | 1.4 | Observed v Predicted Values | 62 |

| 2 | GEN | ERAL | CONSIDERATIONS FOR DATA ANALYSIS | 62 |
|-----|--------|-------|----------------------------------|----|
| | 2.1 | Deriv | ved and transformed data | 62 |
| | 2.2 | Sumr | mary data | 62 |
| 3 | PAR | AMET | ER DEFINITIONS | 63 |
| | 3.1 | Plasn | na Parameters | 63 |
| | | 3.1.1 | Single Dose | 63 |
| | | 3.1.2 | Multiple Dose | 65 |
| API | PENDIX | C: SA | MPLE PAGE LAYOUT | 70 |

#### 1 List of abbreviations

Terminal rate constant  $\lambda_z$ **ALT** Alanine Aminotransferase AP Alkaline Phosphatase Activated Partial Thromboplastin Time **aPTT** Serum Aspartate aminotransferase **AST** Adverse Event AE **AUC** Area under concentration-time curve AUC<sub>t</sub> AUC from time zero to time t AUC<sub>t</sub>/Dose AUC from time zero t to time t, corrected for dose AUC from time zero t to time t, corrected for dose and body weight AUC<sub>t.norm</sub> AUC from time zero to last measurable concentration **AUC**<sub>last</sub> AUC<sub>last</sub>/Dose AUC from time zero to last measurable concentration, corrected for dose AUC from time zero to last measurable concentration, corrected for dose and AUC<sub>last.norm</sub> body weight Twice daily dosing **BID Body Mass Index BMI** BP **Blood Pressure** Below the limit of quantification BOL Confidence Interval CI CK Creatine Kinase CLss/F Apparent Total body clearance at steady state Maximum Plasma Concentration  $C_{max}$ C<sub>max</sub>/Dose C<sub>max</sub> corrected by dose Cmax corrected by dose and body weight C<sub>max,norm</sub> Maximum plasma concentration at steady state  $C_{\text{max.ss}}$ C<sub>max,ss</sub>/Dose Cmax corrected by dose at steady state C<sub>max</sub> corrected by dose and body weight at steady state  $C_{\text{max,ss,norm}}$ Trough Concentration Ctrough Case Report Form **CRF** Clinical StudyReport **CSR** Electrocardiogram **ECG** GLDH Glutamate Dehydrogenase **GGT** Gamma-Glutamyl Transpeptidase Glycated Haemoglobin HbA1C **HMR** Hammersmith Medicines Research HR Heart Rate International Conference on Harmonization **ICH** Investigational Medicine Product **IMP** Liquid Service Formulation **LSF** Lactate Dehydrogenase LDH Mean Corpuscular Haemoglobin **MCH** Mean Corpuscular Haemoglobin Concentration **MCHC MCV** Mean Corpuscular Volume Medical Dictionary for Regulatory Activities MedDR A **MRT** Mean residence time **MRT**inf Mean residence time from time zero to infinity Mean residence time from time zero to last measurable concentration MRT<sub>last</sub>

| N | Number of subjects |
|---|---|
| n | Number of observations used in analysis |
| OD | Once daily dosing |
| OGTT | Oral Glucose Tolerance Test |
| PCI | Potential clinical importance |
| PD | Pharmacodynamic(s) |
| PK | Pharmacokinetic(s) |
| PR | Portion of the ECG from the beginning of the P wave to the beginning of the |
| 1 K | QRS complex, representing attrioventricular node function. |
| PT | Prothrombin Time |
| | Lower quartile |
| Q1 | • |
| Q3 | Upper quartile The ORS complex of the ECC reflects the regid depolarization of the right |
| QRS | The QRS complex of the ECG reflects the rapid depolarization of the right and left ventricles. |
| QT | Portion of the ECG between the onset of the Q wave and the end of the T |
| | wave, representing the total time for ventricular depolarization and |
| | repolarization. |
| QTc | Corrected portion of the ECG between the onset of the Q wave and the end |
| - | of the T wave, representing the total time for ventricular depolarization and |
| | repolarization. |
| QTcB | QTc interval with Bazett's correction method |
| QTcF | QTc interval with Fridericia's correction method |
| R | Accumulation Ratio |
| RBC | Red Blood Cells |
| $R_{ac}C_{max}$ | Accumulation Ratio for C <sub>max</sub> |
| $R_{ac}AUC$ | Accumulation Ratio for AUC |
| RR | Portion of the ECG between consecutive R waves, representing the |
| | ventricular rate |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| t <sub>1/2</sub> | Terminal elimination half-life |
| t <sub>1/2, 0-t</sub> | Dominant half-life |
| TEAE | Treatment-Emergent Adverse Event |
| TSH | Thyroid-Stimulating Hormone |
| t <sub>max</sub> | Time to maximum plasma concentration |
| Vz/F | Apparent Volume of Distribution |
| WBC | White Blood cell |
| WHO | World Health Organisation |
| | <b>5</b> |

### 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:

Helen Topping
Senior Statistician, HMR

Signature

Dr Jeremy Dennison
Principal Investigator, HMR

Signature

Jean-Yves Gillon
Head of Translation, DNDi

Frédéric Monnot
Filarial Team Leader, DNDi

Signature

Principal Investigator, HMR

Signature

Jan-Yves Gillon
Bignature

Jan-Yves Gillon
Date

Prédéric Monnot
Filarial Team Leader, DNDi

Signature

Prédéric Monnot
Filarial Team Leader, DNDi

Signature

Prédéric Monnot
Filarial Program, DNDi

Signature

Principal Investigator, HMR

Signature

Date

Prédéric Monnot
Filarial Team Leader, DNDi

Signature

Prédéric Monnot
Filarial Program, DNDi

Signature

Principal Investigator, HMR

Date

Prédéric Monnot
Filarial Program, DNDi

Signature

Prédéric Monnot
Filarial Program, DNDi

Signature

Prédéric Monnot
Filarial Program, DNDi

#### 3 Introduction

This Statistical Analysis Plan (SAP) is based on the current trial protocol (version 5, 25 July 2018). Where statistical methods differ substantially between this SAP and the protocol, that will be identified in this document.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected during the trial.

The randomisation code will not be broken before this SAP is finalised. If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical study report (CSR). Any deviations from this SAP will be documented in the CSR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Pharmacokinetic analysis will be done using WinNonlin v7 on a Windows PC. Statistical analysis will be done using SAS® 9.3 on a Windows PC.

# 4 Study Objective(s) and Endpoint(s)

# 4.1 Study Objective(s)

#### 4.1.1 Primary Objective(s)

 To investigate the safety and tolerability of emodepside (BAY44-4400) after multiple doses, administered as a LSF oral solution, in healthy male Caucasian subjects.

#### 4.1.2 Secondary Objective(s)

- To investigate the pharmacokinetics (PK) of emodepside (BAY44-4400) after multiple doses, administered as an LSF oral solution.
- To investigate the time-matched profiles of selected pharmacodynamic (PD) markers in plasma, after multiple doses of emodepside (BAY44-4400),

administered as an LSF oral solution.

### 4.2 Study Endpoint(s)

#### 4.2.1 Primary Endpoint(s)

- Adverse events (AEs)
- Physical examination findings
- Neurological examination findings (including assessments of tremor of the hands and fingers, coordination/cerebellar function (finger to finger, finger to nose, with eyes open and closed), pupil size and reaction to light)
- Vital signs: heart rate (HR), systolic and diastolic blood pressure (BP)
- 12-lead ECG (including heart rate (HR), PR, QRS, QTcB, QTcF)
- Clinical laboratory tests:
  - Haematology: haemoglobin, haematocrit, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), platelets, reticulocytes, white blood cells (WBC) including differential, red blood cells (RBC), glycated haemoglobin (HbA1C; at screening only);
  - Coagulation: activated partial thromboplastin time (aPTT), prothrombin time (PT);
  - Biochemistry: serum aspartate aminotransferase (AST), alanine
    aminotransferase (ALT), alkaline phosphatase (AP), glutamate dehydrogenase
    (GLDH), gamma-glutamyl transpeptidase (GGT), lactate dehydrogenase
    (LDH), creatine kinase (CK), amylase, lipase, free T3 and T4, thyroidstimulating hormone (TSH), glucose, cholesterol (HDL, LDL, total),
    triglycerides, creatinine, urea, uric acid, bilirubin (total and conjugated), total
    protein, sodium, potassium, calcium, chloride, and magnesium;
  - At baseline (screening visit 1) and Day 9 additional hormones: leptin and prolactin levels
  - Urinalysis: by dipstick glucose, ketone bodies, specific gravity, occult blood, pH, proteins, leucocytes, bilirubin, urobilinogen, nitrites.
- Ophthalmology assessments: including visual symptoms, past ocular history, best corrected distance visual acuity, colour vision assessment, Amsler grid assessment

#### 4.2.2 Secondary Endpoint(s)

#### Pharmacokinetic Variables:

Emodepside plasma concentration—time data will be used to derive the following PK parameters of emodepside:

• After the first dose of emodepside (Day 0):

- Main PK parameters:
- Cohorts 1 & 2: AUC<sub>24</sub>, AUC<sub>24</sub>/D, C<sub>max</sub>, C<sub>max</sub>/D
- Cohort 3: AUC<sub>12</sub>, AUC<sub>12</sub>/D, C<sub>max</sub>, C<sub>max</sub>/D
- After multiple doses of emodepside (Day 9):
  - Main PK parameters:
  - Cohorts 1 & 2: AUC<sub>∞</sub>, AUC<sub>∞</sub>/D, AUC<sub>24</sub>, AUC<sub>24</sub>/D, C<sub>max,ss</sub>, C<sub>max,ss</sub>/D
  - Cohort 3: AUC∞, AUC∞/D, AUC12, AUC12/D, Cmax,ss, Cmax,ss/D
- Accumulation ratios RA(C<sub>max</sub>) and RA(AUC<sub>tau</sub>) will be calculated
- C<sub>trough</sub> will be derived from the concentration data (Days 1–9).

The above parameters may be calculated for the metabolites of emodepside, as appropriate.

### Pharmacodynamic Variables:

- Time-matched profiles of glucose, glucagon, insulin, and cortisol
- Oral glucose tolerance test (OGTT)

#### **Exploratory PK variables:**

Emodepside plasma concentration—time data will be used to derive the following PK parameters of emodepside:

- After a single dose of emodepside (Day 0):
  - o Cohorts 1 & 2: AUC<sub>24,norm</sub>, C<sub>max,norm</sub>, t<sub>max</sub>, MRT<sub>last</sub>, V<sub>z</sub>/F
  - o Cohorts 3: AUC<sub>12,norm</sub>, C<sub>max,norm</sub>, t<sub>max</sub>, MRT<sub>last</sub>, V<sub>z</sub>/F
- After multiple doses of emodepside (Day 9):
  - AUC<sub>∞,norm</sub>, AUC<sub>12,norm</sub>, AUC<sub>24,norm</sub>, AUC<sub>last</sub>, AUC<sub>last</sub>/D, AUC<sub>last,norm</sub>, C<sub>max,ss,norm</sub>, t<sub>1/2</sub>, λ<sub>z</sub>, t<sub>max</sub>, MRT<sub>∞</sub>, V<sub>z</sub>/F, CL<sub>ss</sub>/F
  - Other optional parameters: AUC<sub>t-inf</sub>, %AUC<sub>extra</sub>, points terminal

### 4.3 Statistical Hypotheses

Except for the analysis of pharmacokinetic data, no formal statistical testing will be done.

# 5 Study Design

This will be a single-centre, single-blind, randomized, placebo-controlled, parallel-group, multiple-dose, dose-escalation study.

Each cohort will comprise 8 healthy Caucasian male subjects, 6 of whom will be randomised to receive emodepside, and 2 of whom will be randomised to receive placebo. 3 cohorts will be recruited, to test 3 multiple dose levels of emodepside LSF oral solution over 10 days.

# 6 Time and Events Table

| | Scre | ening | | | ×(tt- | | | | Day | (s) | | | | | | Long-term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day -28 to -3 | | | | | | | | | | | | | | Follow-up | follow-up<br>visits |
| Procedure | Visit 1 | Visit 2 | -3 | -2 | -1 | 0 | 1 | 2–8 | 9 | 10–14 | 17<br>(±2) | 20<br>(±2) | 23<br>(±2) | 27<br>(±2) | (Day 30<br>±2 Days) | (Days 60,<br>90, and 120<br>±2 Days) <sup>18</sup> |
| Subject demographics and informed consent | Х | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | Х | | | | | × | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Inpatient stay | | | $\leftarrow$ | | | | | | | $\longrightarrow$ | | | | | | X |
| Outpatient visit | X | X | | | | | | | | | X | X | X | X | X | X |
| Drugs of abuse screen and alcohol breath test <sup>1</sup> | Х | | X | | | | | | | | | | | | | × |
| Full physical examination <sup>2</sup> | Х | | | | | | | Х | | X | | | | | X | |
| Short physical examination <sup>2</sup> | | | | | × | Х | Х | х | х | х | Х | Х | Х | Х | | х |
| Full neurological examination <sup>3</sup> | Х | | | | | х | | | | х | | | | | | |
| Short neurological examination <sup>4</sup> | | | | | X | Х | Х | Х | X | Х | Х | Х | х | X | Х | Х |
| Ophthalmological examination <sup>5</sup> | Х | Х | | | | | | | | X | | | | | | |
| Oral Glucose Tolerance<br>Test (OGTT) <sup>6</sup> | | | | Х | | | X | Х | | | | | | | | Х |
| Glucose, insulin, glucagon and cortisol <sup>7</sup> | | | | | X | Х | Х | | X | х | | | | | X | |
| Administration of emodepside <sup>8</sup> | | | | | | Х | Х | х | х | | | | | | | |

HMR code: 16-021

Sponsor code: DNDI-EMO-02

| | Scre | ening | | | | | | | Day | (s) | | | | | | Long-term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | 28 to -3<br>Visit 2 | -3 | -2 | -1 | 0 | 1 | 2–8 | 9 | 10–14 | 17<br>(±2) | 20<br>(±2) | 23<br>(±2) | 27<br>(±2) | Follow-up<br>(Day 30<br>±2 Days) | follow-up<br>visits<br>(Days 60,<br>90, and 120<br>±2 Days) <sup>18</sup> |
| 12-lead safety ECGs9 | X | | | | X | X | X | X | X | X | | | | | X | |
| Vital signs <sup>10</sup> | Х | | | | X | X | X | X | Х | X | X | Х | X | X | X | Х |
| AE monitoring <sup>11</sup> | $\leftarrow$ | | | | | | | | | | | | | | | $\longrightarrow$ |
| PK of emodepside in plasma <sup>12</sup> | | | | | | × | Х | Х | X | Х | Х | х | Х | Х | Х | |
| PK of metabolites of emodepside in plasma <sup>13</sup> | | | | | | х | | | X | | | | | | | |
| PK of emodepside and metabolites in urine <sup>14</sup> | | | | | | x | | | X | | | | | | | |
| Laboratory safety tests <sup>15</sup> | X | | | | Х | Х | Х | X | X | X | | | X | | X | X |
| Serology <sup>16</sup> | Х | | | | | | | | | | | | | | | |
| Leptin and prolactin <sup>7,17</sup> | X | | | | | | | | X | | | | | | | |

- 1. Alcohol breath tests and drugs of abuse screen will be performed at Screening Visit 1 and Day-3. At long-term follow-up visits (Days 60, 90 and 120), only alcohol breath tests will be performed.
- 2. A full physical examination will be done at Screening Visit 1 and Follow-up and before the morning dose on Days 3–8 inclusive, and on Day 14. To include height at Screening Visit 1 and weight at Screening Visit 1 and on the morning of Day –1. Short physical examinations will be done at the following time points:
  - on Day -1: at -24, -23, -22, -20 and -12 h before the morning dose on Day 0
  - on Day 0: before and at 1, 2, 4, and 12 h after the morning dose
  - on Days 1 & 2: before the morning dose
  - on Day 9: before and at the following times after the morning dose: 0.5, 1, 2, 4, 12, 24 h (Day 10), 48 h (Day 11), 72 h (Day 12) and 96 h (Day 13)
  - at outpatients visits on Days 17, 20, 23, 27, and at long-term follow-up visits (Days 60, 90 and 120) (± 2 days)
- 3. A full neurological examination will be done at screening Visit 1, before the morning dose on Day 0 and on Day 14 after the morning dose (120 h).
- 4. A short neurological examination will be given at the following time points:
  - on Day -1: at -24, -23, -22, -20, and -12 h before the morning dose on Day 0
  - on Day 0: at 1, 2, 4, and 12 h after the morning dose
  - on Days 1–8: before the morning dose
  - on Day 9: before and at the following times after the morning dose: 1, 2, 4, 12, 24 (Day 10), 48 (Day 11), 72 (Day 12) and at 96 h (Day 13)
  - at outpatient visits on Days 17, 20, 23, 27 and at Follow-up (Day 30 ± 2 days), and long-term follow-up visits (Days 60, 90 and 120 ±2 days)

HMR code: 16-021

Sponsor code: DNDI-EMO-02

- 5. Ophthalmological examination will be performed at the second screening visit after all other eligibility criteria have been met, and on Day 10. If deemed necessary by the ophthalmologist, additional ophthalmology follow-up visit(s) may be scheduled for eye-related AEs. Subjects will be given the Ishihara test at screening visit 1.
- 6. Blood samples taken for glucose and insulin measurement will be used to complete an Oral Glucose Tolerance Test (OGTT). Samples taken will be:
  - on Day -2: at -48, -47, -46 and -44 h before the morning dose on Day 0
  - on Day 1: before and at 1, 2 and 4 h after the morning dose
  - on Day 8: before and at 1, 2 and 4 h after the morning dose
  - On day 120 at 0, 1, 2 and 4 h time points relative to dosing

Subjects will fast until completion of the OGTT test; lunch will be provided immediately afterwards

- 7. Blood samples for measurement of glucose, insulin, glucagon and cortisol will be taken:
  - on Day -1: at -24, -23, -22, -20 and -12 h before the morning dose on Day 0
  - on Day 0: before and at 1, 2, 4 and 12 h after the morning dose
  - on Day 1: before the morning dose
  - on Day 9: before and at the following time points after the morning dose: 1, 2, 4, 12, 24 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14); and at follow up (Day 30 (± 2 days)). Subjects will fast for the Day 11, 12, 13,14 and 30 time points.

Leptin and prolactin will also be measured at Screening Visit 1 and Day 9, as part of the insulin blood sample.

- 8. Administration of the study medicine will be done in fasting conditions on Days 0-9 at approximatively the same time each morning (±15 mins):
  - in Cohorts 1 & 2, emodepside will be giving in the morning only
  - in Cohort 3, emodepside will be given in the morning and evening (at 12 h intervals). On the last day (day 9), emodepside will be given only in the morning
- 9. 12-lead ECGs will be recorded in triplicate (with 1 minute between recordings) at -24 h (Day -1) before the morning dose on Days 0 and 9; single recordings will be made at all other time points. ECGs will be recorded:
  - at Screening Visit 1 and at Follow-up (Day 30 ± 2 days)
  - on Day -1: at -24, -23.5, -23, -22.5, -22, -21, -20, -16 and -12 h before the morning dose on Day 0
  - on Day 0: before and at 0.5, 1, 1.5, 2, 3, 4, 8 and 12 h after the morning dose
  - on Days 1–8: before the morning dose
  - on Day 9: before and at the following times after the morning dose: 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24 (Day 10), 72 (Day 12) and 120 h (Day 14) after the Day 9 dose

Subjects should rest in the supine position for 10 minutes before ECG measurements.

- 10. Vital signs will comprise blood pressure (BP) and heart rate (HR) at all time points, with oral temperature included at screening and –24 h before the morning dose on Day 0 (Day –1). Subjects should rest in the supine position for 10 minutes before single BP and HR measurements are taken. Vital signs will be measured:
  - at the first screening visit and at Follow-up (Day 30 ± 2 days)
  - on Day -1: at -24, -23.5, -23, -22.5, -22, -21, -20, -16 and -12 h before the morning dose on Day 0
  - on Day 0: before and at 0.5, 1, 1.5, 2, 3, 4, 8 and 12 h after the morning dose
  - on Days 1–8: before the morning dose

HMR code: 16-021

Sponsor code: DNDI-EMO-02

- on Day 9: before and at the following times after the morning dose: 0.5, 1, 1.5, 2, 3, 4, 8,12, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14)
- at outpatients visits on Days 17, 20, 23 and 27 (± 2 days), and long-term follow-up visits (Days 60, 90 and 120 ±2 days)
- 11. Adverse event monitoring will be done throughout the study, but scheduled questioning will be done at the following time points:
  - at Screening Visit 1 and at Follow-up (Day 30 ± 2 days)
  - on Day -1, at -24, -23, -22, -21, -20, -18, -16, -12 h before the morning dose on Day 0
  - on Day 0: before and at 1, 2, 3, 4, 6, 8 and 12 h after the morning dose
  - on Days 1-8: before the morning dose
  - on Day 9: before and at the following times after the morning dose: 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14)
  - at outpatients visits on Days 17, 20, 23 and 27 (± 2 days), and long-term follow-up visits (Days 60, 90 and 120 ±2 days)
- 12. Blood samples for assay of emodepside in plasma will be taken:
  - on Day 0: before and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 h after the morning dose
  - on Days 1-8: before the morning dose
  - on Day 9: before and at the following times after the morning dose: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14)
  - at outpatients visits on Days 17, 20, 23 and 27 (± 2 days), and at Follow-up (Day 30 ± 2 days)

Subjects should rest in the supine position for 10 minutes before blood is drawn (if possible).

- 13. Blood samples for assay of metabolites of emodepside in plasma will be taken:
  - on Day 0: before and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 h after the morning dose
  - on Day 9: before and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 h after the morning dose
- 14. Urine for assay of emodepside and its metabolites may be collected at the following time points:
  - On Day 0: from 0-4, 4-8, 8-12 and 12-24 h after the morning dose
  - On Day 9: from 0-4, 4-8, 8-12 and 12-24 h after the morning dose
- 15. Blood and urine samples for clinical laboratory safety tests (haematology, biochemistry, coagulation & urinalysis) will be taken: at Screening Visit 1; on Day –1 (— 24 h before the morning dose on Day 0); before the morning dose on Days 1, 5 and 8; before, 24 h (Day 10) and 120 h after the morning dose on Day 9 (Day 14); at the Day 23 outpatient visit (± 2 days); at Follow-up (Day 30 ± 2 days); and at long-term follow-up (Days 60, 90 and 120 ± 2 days).
  - Subjects should rest in the supine position for 10 minutes before blood is drawn (if possible).
- 16. Serology tests will comprise HIV 1 & 2, hepatitis B & C, and HbA1c
- 17. Blood samples for measurement of leptin and prolactin will be taken at Screening Visit 1 and before the morning dose on Day 9.
- 18. Subjects will be admitted to the ward on Day 119, before the Day 120 long-term follow-up visit.

### 7 Planned Analyses

### 7.1 Interim Analyses

Interim analyses will be performed. Blinded PK, safety and tolerability data will be reviewed after each cohort for dose selection. Details are given in the Interim Review Plan and in the safety Review Group Charter signed at the beginning of the study.

An additional interim analysis (including interim database lock) will be performed after Cohorts 1 and 2 have completed and unblinded, to evaluate the progression into later phase studies.

#### 7.1.1 Persons responsible for analysis

Stephen Sah (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

### 7.2 Final Analysis

This study will have one database, however Cohorts 1 and 2 will be analysed and reported separately from Cohort 3. Each cohort (Cohorts 1 and 2) and (Cohort 3) will be locked once all subjects have completed, data have been entered, all queries resolved and protocol deviations identified for that cohort of the study. Each cohort (Cohorts 1 and 2) and (Cohort 3) of the study will be unblinded following database lock. Final analyses will be carried out following database lock and unblinding for each cohort (Cohorts 1 and 2) and (Cohort 3) of the study.

#### 7.2.1 Persons responsible for analysis

Helen Topping (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

Duyen Unsworth (HMR) Data Manager

### 8 Sample Size Considerations

### 8.1 Sample Size Assumptions

No formal statistical sample size estimation has been performed, due to the exploratory nature of this study. 6 subjects per dose level (cohort) is considered sufficient to examine the safety and tolerability of emodepside, as well as the pharmacokinetics after single and multiple doses.

### 9 Analysis Populations

The following populations will be identified:

Safety Population: All subjects who received at least one dose of IMP.

PK Concentration Population: All subjects who received at least one dose of IMP and for

whom a pharmacokinetic sample was analysed.

PK Parameter Population: All subjects in the PK Concentration Population for whom

pharmacokinetic parameters can be derived.

In all populations, treatment will be assigned based upon the treatment subjects actually receive regardless of the treatment to which they were randomised.

The primary endpoint will be analysed using the safety population.

#### 9.1 Analysis Datasets

All analysis datasets will be based on observed data, except as outlined in Section 12.2.

### 10 Treatment Comparisons

The treatment comparison of interest is active (emodepside) versus placebo.

# 11 General Considerations for Data Analyses

### 11.1 Data Display Treatment and Other Subgroup Descriptors

The sort order for treatment groups will be placebo, then study treatment in ascending dose order. When a total column is included, it immediately follows the treatment groups which it aggregates.

Listings of data will be sorted and displayed by treatment group, subject number, and also by date and time if applicable.

The treatment descriptions to be used on all tables and listings are:

Treatment GroupsShort DescriptionPlacebo [OD or BID]PLA [OD or BID]Emodepside xx mg [OD or BID]xx mg [OD or BID]

### 11.2 Conventions for Summary Statistics and Data Displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error), median, minimum, and maximum. 95% confidence intervals will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters less than 100 and as integers for values more than 99). The mean and percentiles (e.g. median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

# 12 Data Handling Conventions

# 12.1 Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 12.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (i.e. hours and/or minutes) for adverse events or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (e.g. AE start time from last study medication) will be listed as missing.

Conventions for handling missing plasma concentrations are given in Appendix B.

#### 12.2 Derived and Transformed Data

Baseline will be considered to be the latest value obtained before study drug administration. (e.g. Day 0, pre-dose; or Day -1 if not recorded pre-dose; or Day -2 if not recorded elsewhere etc.)

Laboratory data will be reported in standard units. Out-of-range laboratory tests may be repeated. If a test is out-of-range at a baseline time point and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

Triplicate ECG measurements will be taken at -24 h on Day -1, and at pre dose on Days 0 and 9. The mean of the three measurements taken on Day 0 pre dose for each subject will be used as their baseline value. Single measurements will be made at all other time points.

The pharmacokinetic parameters to be derived are given in Appendix B.

#### 12.3 Assessment Windows

No assessment windows are defined for this report.

### 12.4 Values of Potential Clinical Importance

Any laboratory value outside the reference interval for that variable will be flagged with an 'H' if it is higher than the reference interval, and with an 'L' if it is lower. Additionally, if, during the course of the trial, a variable changes from baseline (Day 0 pre dose) by more than a predetermined amount (as defined by the Principal Investigator, Appendix A), that value will receive a flag 'I' if increased, or 'D' if decreased. Therefore, if a value both falls outside the reference interval and alters from the baseline value by more than the predetermined amount, it will attract a double flag and will be considered to be potentially clinically important.

A vital signs result will be considered to be of potential clinical importance if it falls outside the relevant range below:

| Vital Sign | Range |
|------------------------------------------------|------------------|
| Supine/semi-recumbent systolic blood pressure | 85–160 mm Hg |
| Supine/semi-recumbent diastolic blood pressure | 40–90 mm Hg |
| Supine/semi-recumbent heart rate | 35-100 beats/min |
| Respiration rate | 8-20 per min |
| Oral temperature | 35.5–37.8°C |

QT, QTcB or QTcF > 450 msec and increases in QT, QTcB or QTcF from baseline of > 30 msec will be considered to be potentially clinically important.

# 13 Study Population

### 13.1 Disposition of Subjects

The disposition of all subjects in the safety population will be summarised including number of subjects randomised, number completing the study by treatment, and number withdrawn from the study.

All subjects who withdraw or are withdrawn from the study will be listed by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 13.2 Protocol Deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date.
- Had their treatment assignment unblinded.

In addition, subjects with minor time deviations (measurements taken outside the allowable windows) will be identified. Allowable time windows for pharmacokinetic samples and other procedures are given in section 8.4 of the study protocol.

### 13.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics (e.g. physical examination, vital signs and ECGs) will be listed and summarised.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded using version September 2017 of the World Health Organisation (WHO) Drug Global dictionary.

#### 13.4 Treatment Compliance

Dates and times of dosing will be listed.

### 14 Safety Analyses

Summaries and listings of safety data will use the safety population.

#### 14.1 Extent of Exposure

The dates and times of treatment dosing will be listed to indicate exposure to the study medication.

#### 14.2 Adverse Events

Adverse events will be coded using the version 21.0 or higher of the Medical Dictionary for Regulatory Activities (MedDRA).

All adverse events will be listed.

The number of subjects with at least one treatment-emergent adverse event (TEAE) will be tabulated by actual treatment and MedDRA system organ class. A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pretreatment or having worsened relative to pre-treatment.

For each of the following, the number of adverse events and the number of subjects with adverse events will be summarised:

- TEAEs by system organ class and preferred term
- TEAEs by system organ class, preferred term and severity
- Drug-related ("related" as recorded by the Investigator) TEAEs by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at the greatest severity or causality, for each system organ class/preferred term. Multiple TEAEs in a subject will be counted once per system organ class and preferred term. Adverse events with missing severity and/or causality will be treated as severe and related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

# 14.3 Deaths, Serious Adverse Events and Other Significant Adverse Events

Deaths and serious adverse events will be listed separately (fatal events separate from non-fatal events). Other significant adverse events, as identified by the investigator in the CRF, will be listed separately.

### 14.4 Adverse Events Leading to Withdrawal from the Study

Adverse events leading to withdrawal will be listed separately.

### 14.5 Clinical Laboratory Evaluations

Data from haematology, clinical chemistry, coagulation and urinalysis will be summarised by treatment.

Urinalysis parameters will also be listed.

All laboratory values of potential clinical importance will be listed and all related laboratory results (i.e. haematology, coagulation or clinical chemistry) for subjects with values of potential clinical importance will be listed, separately. Frequencies of laboratory values of potential clinical importance will be summarised.

#### 14.6 Other Safety Measures

#### 14.6.1 Vital signs

Vital signs at each planned assessment, and change in vital signs from baseline at each planned post-baseline assessment, will be summarised by treatment.

Vital signs data of potential clinical importance will be listed.

#### 14.6.2 ECG

QT interval data will be presented using Bazett's (QTcB) and Fridericia's (QTcF) corrections.

ECG data will be summarised by treatment and time point. Differences from baseline (Day 0 pre dose) will be summarised by treatment and time point.

The number of subjects with a potentially clinically important ECG value will be summarised by actual treatment and time point, giving the numbers of subjects with QT, QTcB or QTcF > 450 msec, > 480 msec and > 500 msec, and the numbers of subjects with increases in QT, QTcB or QTcF from baseline of > 30 msec and > 60 msec<sup>3</sup>. A supporting listing of all subjects with an ECG value of potential clinical importance and a separate listing of ECG findings classified as abnormal by the Investigator will also be provided.

#### 14.6.3 Physical examination

Abnormal physical examination findings will be listed.

#### 14.6.4 Neurological examination

Abnormal neurological examination findings will be listed.

#### 14.6.5 Ophthalmology examination

Abnormal ophthalmology examination findings will be listed.

### 15 Pharmacokinetic Analyses

Analytical Services International Ltd will measure the plasma concentrations of emodepside. The pharmacokinetic analysis will be done by Statistics and Data Management Department at HMR. Pharmacokinetic parameters will be calculated using WinNonlin, version 7.0 or higher.

The pharmacokinetic parameters to be derived are given in Appendix B.

PK concentration data will be summarised using the PK concentration population. PK parameters will be summarised using the PK parameter population.

For log normally distributed parameters, the primary measure of central tendency will be the geometric mean<sup>4</sup>; for other parameters, it will be the arithmetic mean or median.

For all variables N (number of subjects receiving the treatment/formulation in the population), n (number of observations), arithmetic mean, median, minimum, maximum, SD, %CV, and the 95% confidence interval for the arithmetic mean will be provided. For log-transformed variables, all of the above plus the geometric mean, which is the anti-logged arithmetic mean of log-transformed variables, its 95% confidence interval and the SD of the logs will be provided.

The between-subject CV will be calculated using:

1. %CVb = 100 \* (SD/Mean) with SD and Mean of untransformed data

2.  $\%CVb = 100 * \sqrt{(exp(SD)^2 - 1)}$  with SD of log-transformed data

#### 15.1 Plasma PK

#### 15.1.1 Pharmacokinetic Concentration Data

The plasma concentrations of emodepside and metabolites (if applicable) will be listed and summarised by treatment.

Using actual sample times, linear and semi-logarithmic concentration-time plots of each analyte for each subject will be prepared. For subjects receiving more than one dose of a treatment, profiles will be included for all doses on the same plot. The same linear and logarithmic scales will be used for each subject. The linear and semi-logarithmic plots for a given subject will be presented on the same page. For clarity in presentation, individual profiles for different analytes will generally be separate.

Nominal blood sampling times will be used to calculate the geometric mean (geo SD) drug concentrations at each time point. Comparative linear and semi-logarithmic plots of the geometric mean (with geo standard deviation error bars) concentration-time data for each group will be prepared.

#### 15.1.2 Pharmacokinetic Parameters

The pharmacokinetic parameters of emodepside and metabolites (if applicable) will be listed and summarised by treatment.

#### 15.2 Urinary PK

If concentrations of emodespide and metabolites (if applicable) in urine are determined, the amount of emodepside excreted in the urine will be estimated and listed.

### 16 Pharmacodynamic Analyses

Summaries and listings will use the safety population.

Pharmacodynamic variables (glucose, insulin, glucagon, cortisol and oral glucose tolerance test) at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by treatment.

Individual PD subject profiles plotted against time will be presented for both absolute values and change from baseline.

### 17 References

1. International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials - ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.

- 2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.
- International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc
   Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs.
   Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.
- 4. Julious, SA & Debarnot, CAM (2000) "Why are Pharmacokinetic Data Summarised by Arithmetic Means?", Journal of Biopharmaceutical Statistics, 10 (1), p55-71

#### 18 ATTACHMENTS

### 18.1 Table of Contents for Data Display Specifications

For overall page layout refer to Appendix C.

Tables, figures and listings will be labelled A (for Cohorts 1 and 2) and B (for Cohort 3), e.g. 14.1A, 14.1B. Separate tables will be produced for Cohorts 1 and 2 and for Cohort 3.

The numbering in the tables below will take precedence over the numbering in the shells.

The following tables and figures will be produced (templates provided in Section 18.2.1):

| Table | Description | Population | Source<br>Listing | Template<br>(Shells<br>below) |
|---|---|---|---|---|
| 10.1 | Summary of subject disposition | Safety | 16.2.1.2, | T_SD1 |
| | | | 16.2.3.1 | |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of demographic characteristics | Safety | 16.2.4.1 | <u>T_DM1</u> |
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1.1 | Summary of emodepside plasma pharmacokinetic concentration-time | PK | 16.2.6.1.1 | T PK1 |
| | data [units] | Concentration | | _ |
| 14.2.1.2 | Summary of derived emodepside plasma pharmacokinetic parameters | PK Parameter | 16.2.6.1.2 | <u>T PK3</u> |
| 14.2.1.3 | Summary of log-transformed derived emodepside plasma | PK Parameter | 16.2.6.1.2 | T_PK4 |
| | pharmacokinetic parameter | | | _ |
| 14.2.2.1 | Summary of glucose | Safety | 16.2.6.2.1 | <u>T_LB2</u> |
| 14.2.2.2 | Summary of insulin | Safety | 16.2.6.2.1 | T_LB2 |
| 14.2.2.3 | Summary of glucagon | Safety | 16.2.6.2.1 | T_LB2 |
| 14.2.2.4 | Summary of cortisol | Safety | 16.2.6.2.1 | <u>T_LB2</u> |
| 14.2.3.1 | Summary of oral glucose tolerance test results | Safety | 16.2.6.2.1 | <u>T_LB2</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of treatment-emergent adverse events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.1.2 | Summary of drug-related treatment-emergent adverse events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.1.3 | Summary of treatment-emergent adverse events by severity | Safety | 16.2.7.1 | <u>T_AE3</u> |
| 14.3.2.1 | Listing of fatal adverse events | Safety | 16.2.7.1 | L AE1 PC |
| 14.3.2.2 | Listing of non-fatal serious adverse events | Safety | 16.2.7.1 | L_AE1_PC |
| 14.3.2.3 | Listing of other significant adverse events | Safety | 16.2.7.1 | L AE1 PO |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | | - |
| 14.3.4 | Summary of laboratory values of potential clinical importance | Safety | 16.2.8.1, | T_LB1 |
| 14.3.5.1 | Summary of chemistry laboratory values | Safety | 16.2.8.3<br>16.4 | T LB2 |
| 14.3.5.1 | Summary of haematology laboratory values | Safety | 16.4 | T LB2 |
| 14.3.5.3 | Summary of nacinatology laboratory values | Safety | 16.4 | T LB2 |
| 14.3.5.4 | Summary of urinalysis results | Safety | 16.2.8.5 | <u>T_LD2</u><br>T_UR1 |

| Table | Description | Population | Source<br>Listing | Template<br>(Shells<br>below) |
|---|---|---|---|---|
| 14.3.6.1 | Summary of vital signs | Safety | 16.4 | <u>T_VS1</u> |
| 14.3.7.1 | Summary of ECG values | Safety | 16.4 | T EG2 |
| 14.3.7.2 | Summary of ECG values and changes in ECG values of potential clinical importance | Safety | 16.2.9.2 | T_EG3 |

| Figure | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1.1 | Individual emodepside plasma concentration-time plots (linear and semi-log) | PK<br>Concentration | 16.2.6.1.1 | <u>F_PK1</u> |
| 14.2.1.2 | Geometric mean (with geo SD error bars) emodepside plasma concentration-time plots (linear and semi-log) | PK<br>Concentration | 16.2.6.1.1 | <u>F_PK2</u> |
| 14.2.2.1 | Individual glucose-time plots | Safety | 16.4 | F_SAF1 |
| 14.2.2.2 | Individual insulin-time plots | Safety | 16.4 | F_SAF1 |
| 14.2.2.3 | Individual glucagon-time plots | Safety | 16.4 | F_SAF1 |
| 14.2.2.4 | Individual cortisol-time plots | Safety | 16.4 | <u>F_SAF1</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1 | Individual systolic blood pressure-time plots | Safety | 16.4 | F SAF1 |
| 14.3.2 | Individual diastolic blood pressure-time plots | Safety | 16.4 | F_SAF1 |
| 14.3.3 | Individual heart rate-time plots | Safety | 16.4 | F SAF1 |
| 14.3.4 | Individual QTcF-time plots | Safety | 16.4 | F_SAF1 |
| 14.3.5 | Individual QTcB-time plots | Safety | 16.4 | F SAF1 |

The following abbreviated listings will be produced (templates provided in Section 18.2.2):

| Listing | Description | Template<br>(Shells<br>below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | |
| 16.2.1.1 | Listing of study dates | L SD1 PG |
| 16.2.1.2 | Listing of reasons for withdrawal | L SD2 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of subjects with inclusion/exclusion criteria deviations | L DV1 PG |
| 16.2.2.2 | Listing of subjects with time deviations | L TD1 PG |
| 16.2.2.3 | Listing of subjects with other protocol deviations | L DV2 PG |
| 16.2.3 | Analysis sets, including subjects excluded from analysis | |
| 16.2.3.1 | Listing of analysis populations | L AN1 PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of demographic characteristics | L DM1 PG |
| 16.2.4.2 | Listing of concomitant medications | L CM1 PG |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of exposure data | L EX1 PG |
| 16.2.6 | Pharmacokinetic and pharmacodynamic data | |
| 16.2.6.1.1 | Listing of emodepside plasma pharmacokinetic concentration-time data | L_PK1_PG |
| 16.2.6.1.2 | Listing of derived emodepside plasma pharmacokinetic parameters | L PK4 PG |
| 16.2.6.1.3 | Listing of emodepside plasma urine sample collections | L PK2 PG |
| 16.2.6.1.4 | Individual emodepside plasma concentration-time plots for estimation of λz, with regression line | <u>F_PK10</u> |
| 16.2.6.2.1 | Listing of PD concentration-time data | L PK1 PG |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of all adverse events | L AE1 PG |
| 16.2.7.2 | Listing of serious adverse events | L AE1 PG |
| 16.2.7.3 | Listing of adverse events leading to withdrawal from study | L AE1 PG |
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of clinical chemistry abnormalities of potential clinical importance | L LB1 PG |
| 16.2.8.2 | Listing of all clinical chemistry laboratory data for subjects with PCI | L LB2 PG |

| Listing | Description | Template<br>(Shells<br>below) |
|---|---|---|
| | abnormalities* | |
| 16.2.8.3 | Listing of haematology abnormalities of potential clinical importance | L LB1 PG |
| 16.2.8.4 | Listing of all haematology laboratory data for subjects with PCI abnormalities* | L LB2 PG |
| 16.2.8.5 | Listing of urinalysis data | <u>L URI PG</u> |
| 16.2.9 | Vital signs, ECG variables and physical findings | |
| 16.2.9.1 | Listing of vital signs of potential clinical importance | L VS1 PG |
| 16.2.9.2 | Listing of ECG values of potential clinical importance | L EG1 PG |
| 16.2.9.3 | Listing of abnormal ECG findings | L EG2 PG |
| 16.2.9.4 | Listing of abnormal physical examination findings | L PE1 PG |
| 16.2.9.5 | Listing of abnormal neurological examination findings | L NE1 PG |
| 16.2.9.6 | Listing of abnormal ophthalmology examination findings | L PE1 PG |

<sup>\*</sup> ICH does not require full listings of lab data so only subjects with double-flagged values will be listed.

Complete listings of all data collected in this study will also be produced.

# 18.2 Data Display Specifications

### 18.2.1 Table Outlines

#### Template T\_SD1

Table 10.1 Summary of subject disposition

| Population | Status | Reason for Withdrawal | Treatment 1<br>(N=xx)<br>n (%) | Treatment 2<br>(N=xx)<br>n (%) | Etc | All Subjects<br>n (%) |
|---|---|---|---|---|---|---|
| Safety | Included | | XX | xx | | xx |
| , | Completed<br>Withdrawn | | xx (xx) | xx (xx) | | xx (xx) |
| | | Death | xx (xx) | xx (xx) | | xx (xx) |
| | | Adverse Events | xx (xx) | xx (xx) | | xx (xx) |
| | | Withdrawal by subject | xx (xx) | xx (xx) | | xx (xx) |
| | | Study terminated by<br>Sponsor | xx (xx) | xx (xx) | | xx (xx) |
| | | Lost to follow-up | xx (xx) | xx (xx) | | xx (xx) |
| | | Other | xx (xx) | xx (xx) | | xx (xx) |
| Alternative 1 (if applicable) | Included | | | | | |
| Alternative 2 (if applicable) | Included | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

#### Template T\_DM1

Table 14.1 Summary of demographic characteristics

| Variable | Statistics | Treatment 1 | Treatment 2 | Etc | All Subjects (N=xx) |
|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | | |
| Age (y) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Gender | Male | | | | |
| Race (%) | American Indian or Alaskan | | | | |
| | Native | | | | |
| | Asian | | | | |
| | Black | | | | |
| | Native Hawaiian or other | | | | |
| | Pacific Islander | | | | |
| | White | | | | |
| | Other | | | | |
| Ethnicity (%) | Hispanic or Latino | | | | |
| | Not Hispanic or Latino | | | | |
| Height (cm) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Weight (kg) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |

| Variable | Statistics | Treatment 1 (N=xx) | Treatment 2<br>(N=xx) | Etc | All Subjects (N=xx) |
|---|---|---|---|---|---|
| | Min | | | | |
| | Max | | | | |
| BMI (kg/m2) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Smoker (%) | n | | | | |
| Cigarettes* | n | | | | |
| (daily) | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Alcohol* | n | | | | |
| (units/week) | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Xanthine* | | | | | |
| (units/week) | | | | | |

<sup>\*</sup>includes only those subjects who smoke/drink alcohol/drink beverages containing Xanthine

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and additional demographic characteristics

#### Template T\_PK1

Table 14.2.xx Summary of emodepside plasma pharmacokinetic concentration-time data [units]

| | {Add.<br>time | Planned<br>Relative | | No. | | 95% CI | | | | | | Geom. | Geom. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | var.} | Time | n | Imputed | Mean | (Lower,Upper) | SD | %CVb | Median | Min | Max | Mean | SD |
| Treatment 1 | | Pre-dose | x | x | хххх.х | (xxxx.x,xxxxxx) | | xx.x | хххх.х | хххх | хххх | | |
| (N=xx) | | 30 min | × | x | xxxx.x | (xxxx.x,xxxx.x) | xx.xx | xx.x | xxxx.x | XXXX | xxxx | | |
| | | 1 hr | x | x | хххх.х | (xxxxxxxxxx) | xx.xx | хх.х | хжж.х | хххх | XXXX | | |
| Treatment 2 | | Pre-dose | x | x | хххх.х | (xxxx.x,xxxxx) | xx.xx | xx.x | xxxx.x | xxxx | xxxx | | |
| (N=xx) | | 30 min | x | x | XXXX.X | (xxxxx,xxxxxx) | xx.xx | xx.x | хххх.х | XXXX | хххх | | |
| | | 1 hr | x | x | xxxx.x | (xxxx.x,xxxx.x) | xx.xx | xx.x | xxxx.x | xxxx | xxxx | | |

Source: Listing 16.2.xx

Programming notes:

Continued with all dose levels and timepoints

#### Template T\_PK3

Table 14.2.xx Summary of derived emodepside plasma pharmacokinetic parameters

| Parameter | Treatment | {Additional time variables} | n | Mean | 95% CI<br>(Lower,Upper) | SD | %CVb | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| AUC <sub>t</sub> (units) | Treatment 1 (N=xx) | | хх | xxxx.xx | (xxxx.xx,xxxx.xx) | хх.ххх | xx.x | xxxx.xx | xxxx.x | XXXX.X |
| | Treatment 2 (N=xx) | | хx | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | xx.x | xxxx.xx | xxxx.x | xxxx.x |
| C <sub>max</sub> (units) | Treatment 1 (N=xx) | | ХX | xxxx.xx | (xxxx.xx,xxxx.xx) | хх.ххх | xx.x | xxxx.xx | xxxx.x | XXXX.X |
| | Treatment 2 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | хх.хх | xx.x | xxxx.xx | xxxx.x | xxxx.x |

Source: Listing 16.2.xx

Programming notes:

Continued with all dose levels, timepoints and parameters

#### Template T\_PK4

Table 14.2.xx Summary of log-transformed derived emodepside plasma pharmacokinetic parameters

| | | {Additional | | | - | | |
|---|---|---|---|---|---|---|---|
| | | time | | Geom | 95% CI | | |
| Parameter | Treatment | variables} | n | Mean | (Lower,Upper) | SD (logs) | %CVb |
| AUC <sub>last</sub> (units) | Treatment 1 (N=xx) | • | | XXXX.XX | (xxxx.xx,xxxxxx) | хх.хх | XX.XX |
| | Treatment 2 (N=xx) | | | XXXX.XX | (xxxx,xxxxxx) | xx.xx | xx.xx |
| C <sub>max</sub> (units) | Treatment 1 (N=xx) | | | xxxx.xx | (xxxx.xx,xxxxxx) | xx.xx | xx.xx |
| | Treatment 2 (N=xx) | | | xxxx.xx | (xxxx.xx,xxxxxxx) | xx.xx | xx.xx |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels, timepoints and parameters

#### Template T\_AE1

Table 14.3.3.xx Summary of treatment-emergent adverse events

| | | Treatment 1 (N=xx) | Treatment 2 (N=xx) | Etc |
|---|---|---|---|---|
| System Organ Class | Preferred Term | n (%) | n (%) | |
| Number of subjects with AEs | | x (xx.x) | x (xx.x) | |
| Gastrointestinal disorders | Total number of subjects | x (xx.x) | x (xx.x) | |
| | Abdominal discomfort | x (xx.x) [xx] | x (xx.x) [xx] | |
| | Abdominal pain<br>↓ | x (xx.x) [xx] | x (xx.x) [xx] | |
| Nervous system disorders | Total number of subjects | | | |
| | Dizziness | | | |
| | Headache | | | |
| | <b>†</b> | | | |
| <b>↓</b> | <b>↓</b> | | | |

n = number of subjects (subjects with ≥1 adverse event are counted only once per system organ class and preferred term)

[] = number of adverse events

Based on MedDRA version xx.x

Source: Listing 16.2.xx

Programming notes:

Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms.
#### Template T\_AE3

Table 14.3.3.xx Summary of treatment-emergent adverse events by severity

| | | Treatment 1 (N=xx) | Treatment 2 (N=xx) | Etc |
|---|---|---|---|---|
| System Organ Class | Preferred Term | n (%) | n (%) | |
| Number of subjects with AEs | | x (xx.x) | x (xx.x) | |
| Gastrointestinal disorders | Abdominal discomfort | x (xx.x) | x (xx.x) | |
| | Abdominal pain | x (xx.x) | x (xx.x) | |
| | <b>†</b> | | | |
| Nervous system disorders | Dizziness | | | |
| | Headache | | | |
| | <b>↓</b> | | | |
| <b>↓</b> | <b>↓</b> | | | |

n = number of subjects (subjects with ≥1 adverse event are counted only once per system organ class and preferred term)

Based on MedDRA version xx.x

Source: Listing 16.2.xx

Programming notes:

Each preferred term counted only once across all severities for each subject/treatment

Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

 ${\it Presented for all applicable MedDRA system organ classes and terms.}$ 

Sponsor code: DNDI-EMO-02

#### Template T\_LB1

Table 14.3.4.xx Summary of laboratory values of potential clinical importance

| | | Planned Relative | | Doub | le Flags |
|---|---|---|---|---|---|
| Laboratory Test (units) | Treatment | Time | n | н | LD |
| | Treatment 1 (N=xx) | | | | |

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Source: Listing 16.2.xx

Programming notes:

Continued with all tests, treatment groups and time points. n = total number of results for that parameter

#### Template T\_LB2

Table 14.3.5.xx Summary of chemistry laboratory values

| | | | | | | | | | | Ch | ange f | rom Baselin | e | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test | | Planned | | | | | | | | | | | | |
| (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes:

Continued with all treatments and time points

Sponsor code: DNDI-EMO-02

#### Template T\_UR1

Table 14.3.5.xx Summary of urinalysis results

| | Planned Relative | e | Treatment 1 | L (N=xx) | Treatment 2 | 2 (N=xx) |
|---|---|---|---|---|---|---|
| Laboratory Test | Time | Result | n | % | n | % |
| <del></del> | Time 1 | Positive | х | х | | |
| | | Negative | х | X | | |
| | | Not Done | x | | | |
| | Time 2 | Positive | | | | |
| | | Negative | | | | |
| | | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes:

Results recorded as received, e.g. Negative, Trace, etc; urine pH summarised as <5, 5-8, >8; specific gravity summarised as <=1.005, 1.006 - 1.010, 1.011 - 1.015, 1.016 - 1.020, 1.021 - 1.025, 1.026 - 1.029, >=1.030. Continued with all treatment groups and time points. The n's sum to N but the calculated percentages exclude Not Done.

#### Template T\_VS1

Table 14.3.6.xx Summary of vital signs

| | | | | | | | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | |
| Variable (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median Min | Max |
| Systolic BP (mmHg) | Treatment 1 (N=xx) | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes:

Continued with all variables, treatments and time points

Sponsor code: DNDI-EMO-02

#### Template T\_EG2

Table 14.3.7.xx Summary of ECG values

| | | | | | | | | | Cl | hange | from Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Planned Relative<br>Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Treatment 1 (N=xx) | | | | | | | | | | | | | |
| Treatment 2 (N=xx) | | | | | | | | | | | | | |
| Treatment 1 (N=xx) | | | | | | | | | | | | | |
| Treatment 2 (N=xx) | | | | | | | | | | | | | |
| | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Planned Relative Treatment Time n Mean SD Median Min Max n Mean Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Planned Relative Treatment Time n Mean SD Median Min Max n Mean SD Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Planned Relative Treatment Time n Mean SD Median Min Max n Mean SD Median Treatment 1 (N=xx) Treatment 2 (N=xx) Treatment 1 (N=xx) | Treatment 1 (N=xx) Treatment 1 (N=xx) Treatment 1 (N=xx) |

Source: Listing 16.2.xx

Programming notes:

Continued with all treatment groups and time points

Do not summarise RR or QRS axis

Template T\_EG3

Table 14.3.7.xx Summary of ECG values and changes in ECG values of potential clinical importance

| | | Planned | | | | | | | >30-6 | 0 msec | >60 | msec |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Relative | 451 – 48 | 30 msec | 481 - 50 | 00 msec | > 500 | msec | Incr | ease | Incr | ease |
| Variable | Treatment | Time | n | % | n | % | n | % | n | % | n | % |
| QT interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| | Treatment 2 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| QTcF interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points. n = total number of results for that parameter

## 18.2.2 Figure Outlines

#### Template F\_PK1

Figure 14.2.xx Individual emodepside plasma concentration-time plots (linear and semi-log)

Subject x Treatment x





Programming notes:

For parallel group studies with a multiple days, page by treatment and include one subject with both days on same page

Template F\_PK2

Figure 14.2.xx Geometric Mean (with Geo SD error bars) emodepside plasma concentration-time plots (linear and semi-log)



BLQ values observed post dose are imputed to half of the LLOQ. Pre dose values are imputed to zero

Programming notes: Offset treatment groups (to both sides of timepoint) to minimise overlapping error bars

Figure 16.2.xx Individual emodepside plasma concentration-time plots for estimation of lambda-z, with regression line



#### Template F\_SAF1

Figure 14.3.1 Individual systolic blood pressure-time plots



Programming note: Plots are by treatment groups Continue with all parameters

Sponsor code: DNDI-EMO-02

### 18.2.3 Listing Outlines

| Template L_ | SD1 | PG |
|-------------|-----|----|
|-------------|-----|----|

Listing 16.2.x.xx Listing of study dates

Final

Treatment Subject Screening First Dose Follow Up

Programming notes: L

Lists dates for screening, each dosing period and follow up

#### Template L\_SD2\_PG

Listing 16.2.x.xx Listing of reasons for withdrawal

Date of Study
Treatment Subject Withdrawal Day Reason

Programming notes:

Reason for withdrawal is concatenation of reason and details

#### Template L\_DV1\_PG

Listing 16.2.x.xx Listing of subjects with inclusion/exclusion criteria deviations

Treatment Subject Type Criterion
Inclusion
Exclusion

Sponsor code: DNDI-EMO-02

#### Template L\_TD1\_PG

Listing 16.2.x.xx Listing of subjects with time deviations

| | | Planned | | Allowed | Actual | Time outside the |
|---|---|---|---|---|---|---|
| | | Relative | | deviation | deviation | deviation window |
| Treatment | Subject | Time | Procedure | (h:min) | (h:min) | (h:min) |

Programming notes:

Only include time deviations which exceed the allowed deviation

#### Template L\_DV2\_PG

Listing 16.2.x.xx Listing of subjects with other protocol deviations

Treatment Subject Protocol Deviation

#### Template L\_AN1\_PG

Listing 16.2.x.xx Listing of analysis populations

Safety

Treatment Subject Population Population 1 Population 2 Etc.

Sponsor code: DNDI-EMO-02

#### Template L\_DM1\_PG

Listing 16.2.x.xx Listing of demographic characteristics

| | | Date of | Age | | | | Height | Weight | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | screening visit | (y) | Gender | Race | Ethnic origin | (cm) | (kg) | BMI (kg/m2) | Etc (units) |
| Treatmer | nt 1 | | | | | | | - | | |
| <b>↓</b> | | | | | | | | | | |

Programming notes:

A by-subject listing of demographic characteristics including:

Treatment

Subject

Date of screening visit

Age

Gender

Race / Ethnic Origin

Height (if collected only once during the study)

Weight (if collected only once during the study)

Smoking History

Alcohol Consumption

Xanthine

Additional study-specific demography characteristics included on the CRF

Sponsor code: DNDI-EMO-02

#### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of concomitant medications

| | | ATC Class/ | Drug Name/ | Dose/ | Date/time Started/ | Time Since Last | Started Pre- | Ongoing |
|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Medication Code* | Indication | Freq/Route | Date Stopped | Dose | Trial? | Medication? |

Coded using WHODrug Global version xx.x\*

Programming notes:

\* only include this column and the footnote if coding used

Include dose and units (e.g. 5 mg)/Freq/Route

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of exposure data

| | | Start Date/ | Stop Date/ | Duration | | Dose | Formulation/ | |
|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Start Time of Dose | Stop Time of Dose | (days) | Dose | Unit | Route | Frequency |
| Treatment 1 | 1001 | 01JAN2002 | 15FEB2002 | 46 | 25 | mg | Tablet/ | 2xday |
| | | 23:59 | 15:30 | | | | Oral | |

#### Template L\_PK1\_PG

Listing 16.2.6.xx Listing of emodepside plasma pharmacokinetic concentration-time data

| | | {Add. | | | | | | Actual Relative | |
|---|---|---|---|---|---|---|---|---|---|
| | | time | | | Planned | Actual time | Time Deviation | Time | |
| Treatment | Subject | var.} | Date | Study Day | <b>Relative Time</b> | (hh:mm) | (min) | ( h) | Concentration (units) |

Below the Limit of Quantification (BLQ) is < xx units (e.g. 1 ng/mL)

Programming notes:

Values below LLOQ are shown as BLQ. Check LLOQ value in final PK spreadsheet for each analyte.

Sponsor code: DNDI-EMO-02

#### Template L\_PK2\_PG

Listing 16.2.6.xx Listing of emodepside urine sample collections

| | | | | | | | | | | ve amount<br>reted |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | {Add.<br>time<br>var.} | Study Day | Planned Relative<br>Time | Start Date/<br>Start Time | Stop Date/<br>Stop Time | Conc. (units)/<br>Volume (units) | Amount<br>excreted<br>(units) | Absolute<br>(units) | Relative<br>to dose<br>(%) |
| | | | | Pre-dose | | | xxx.xx/<br>xxx.xx | ххх.хх | | , , |
| | | | | 0-12 h | | | xxx.xx/<br>xxx.xx | ххх.хх | ххх.хх | x.xx |
| | | | | 12-24 h | | | xxx.xx/<br>xxx.xx | ххх.хх | xxx.xx | x.xx |

Programming notes: Planned relative time is in the form "Oh to 12h" For spot samples (pre dose and follow up) only report urine concentrations and volumes.

#### Template L\_PK4\_PG

Listing 16.2.xx Listing of derived emodepside plasma pharmacokinetic parameters

| | | {Add. | | | | | |
|---|---|---|---|---|---|---|---|
| | | time | AUC <sub>inf</sub> | AUC <sub>t</sub> | $C_{max}$ | t <sub>1/2</sub> | t <sub>max</sub> |
| Treatment | Subject | var.} | (units) | (units) | (units) | (units) | (units) |

Programming notes: Continue with all parameters

Sponsor code: DNDI-EMO-02

#### Template L\_AE1\_PG

Listing 16.2.x.xx Listing of all adverse events

| Treatment | Subject | System Organ Class / Preferred Term/ Verbatim Text | Outcome/ Onset Date/Time/ Resolved Date/Time/ Duration | Time Since Last<br>Dose | Severity/<br>Serious/<br>Withdrawal | Frequency/<br>Action Taken (1)/<br>Other Action<br>Taken | Related to Study Drug/ Treatment Emergent? |
|---|---|---|---|---|---|---|---|
| Treatment 1 | 1001 | Gastrointestinal Disorders /<br>Intestinal Spasm /<br>Entero-spasm | Resolved/<br>24SEP2003 13:05/<br>27OCT2003 7:50/ | 10d 7h 3m | Mild/<br>No/<br>Yes | Intermittent/ Dose<br>not changed/<br>None | Possibly/<br>Yes |
| | | | 34d 4h 5m | | | | |

<sup>(1)</sup> Action Taken with Study Treatment

Programming notes:

For the listing of "other significant AEs" include (from ICH E3) AEs leading to withdrawal, AEs leading to dose reduction (including drug withdrawn, interrupted, reduced or similar) and AEs with AEOSE=Y. If AEOSE has not been collected then use "Otherwise significant" in the CRF.

Sponsor code: DNDI-EMO-02

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of clinical chemistry abnormalities of potential clinical importance

| | | | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Relative | | Study | | | | | Clinically |
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Reference Interval | RI | BL | Significant? |
| Treatment 1 | 1001 | Alk Phos (U/L) | Time 1 | 01JAN2002 | -1 | 64.00 | 32.0 - 92.0 | | | |
| | | | | 13:34 | | | | | | |
| | | | Time 2 | 01APR2002 | 85 | 84.00 | 32.0 - 92.0 | | | |
| | | | | 07:22 | | | | | | |
| | | ALT (U/L) | Time 1 | 01JAN2002 | -1 | 29.00 | 10.0 - 40.0 | | | |
| | | | | 18:56 | | | | | | |
| | | | Time 2 | 01APR2002 | 85 | 70.00 | 10.0- 40.0 | н | i | Υ |
| | | | | 09:22 | | | | | | |

RI for Reference Interval flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes:

Lists only double-flagged subjects

Sponsor code: DNDI-EMO-02

#### Template L\_LB2\_PG

Listing 16.2.x.xx Listing of all clinical chemistry laboratory data for subjects with PCI abnormalities

| | | Planned<br>Relative | | Alkaline Ph | osphatase (IL | J/L) | Alanine A | mino Tra<br>(IU/L) | nsferase | Aspartate | : Amino Trai<br>(IU/L) | nsferase | Total E | Bilirubin (UN | MOL/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | Result | RI | BL | Result | RI | BL | Result | RI | BL | Result | RI | BL |
| | | Planned | | | | | | | | | | | | | |
| | | Relative | | Chlorid | e (MMOL/L) | | Gluce | se (MMC | L/L) | Potas | sium (MMO | L/L) | Sod | ium (MMO | L/L) |
| Treatment | Subject | Time | Date/Time | Result | RI | BL | Result | RI | BL | Result | RI | BL | Result | RI | BL |
| | | | Planned<br>Relative | | Ca | lcium (M | MOL/L) | | Creatinin | ne (UMOL/L) | | | Etc. | | |

RI for Reference Interval flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes:

Lists only double-flagged subjects

Include all parameters for the study following the order from the lab report (above is a guide only)

Sponsor code: DNDI-EMO-02

#### Template L\_URI\_PG

Listing 16.2.x.xx Listing of urinalysis data

| | Planned | | | Specific | Gravity | pН | l | Prote | ein | Gluc | ose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Relative | | | | | | | | | |
| Treatment | Subject | Time | Date/Time | Result | RI | Result | RI | Result | RI | Result | RI |

RI for Reference Interval flag, H = Above reference interval, L = Below reference interval, A = Abnormal result

Programming notes:

Include all parameters for the study following the order from the lab report (above is a guide only)

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of vital signs of potential clinical importance

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | <b>Blood Pressure</b> | <b>Blood Pressure</b> | Etc |
| Treatment | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| | | 24 H | 26SEP2012:09:57 | 63 | 148* | |

<sup>\*</sup> Value of potential clinical importance

Sponsor code: DNDI-EMO-02

Template L\_EG1\_PG

Listing 16.2.x.xx Listing of ECG values of potential clinical importance

| | | | | | | | | QT Int. | (msec) | QTcB | (msec) | QTcF | (msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Heart | | QRS | QRS | | Change | | Change | | Change |
| | | Planned | | Rate | PR Int. | Dur. | Axis | | from | | from | | from |
| Treatment | Subject | Relative Time | Date/Time | (bpm) | (msec) | (msec) | (deg) | Observed | Baseline | Observed | Baseline | Observed | Baseline |
| | | 24 H | 26SEP2012:09:57 | 63 | 148 | 78 | 50 | 390 | 32.7 * | 399 | -27.7 | 396 | -6.5 |

Programming notes:

Do not list RR

<sup>\*</sup> Value of potential clinical importance

Sponsor code: DNDI-EMO-02

#### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of abnormal ECG findings

**Planned Relative** 

Comment on Clinical

Treatment

Subject

Time

Date/Time

ECG Finding

Significance

Programming notes:

Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of abnormal physical examination findings

**Planned Relative** 

Treatment

Subject

Time

Date/Time

Site

Details

**Programming Notes:** 

List only findings with an 'abnormal' result.

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

For ophthalmology listing replace column Site with Test.

Sponsor code: DNDI-EMO-02

Template L\_NE1\_PG

Listing 16.2.x.xx Listing of abnormal neurological examination findings

Planned

Treatment Subject Relative Time Date/Time Type Assessment Details

**Programming Notes:** 

Type = (Mental Status, Cranial Nerves, etc.)

List only findings with an 'abnormal' result.

If subjects have multiple abnormal assessment at a given time, create a separate row for each assessment.

# **Appendix A: Laboratory Ranges**

# Pre-determined Changes for Laboratory Data (from FL140 v4)

| | | | | Delta ranges | |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable decrease | Acceptable increase |
| Activated partial thromboplastin time | APTTT | sec | Both | - 8.0 | + 8.0 |
| Alanine transferase | ALTN | IU/L | F | - | + 30 |
| Alanine transferase | ALTN | IU/L | M | - | + 30 |
| Albumin | ALB | g/L | Both | - 8 | + 8 |
| Alkaline phosphatase | ALPN | IU/L | Both | - 30 | + 30 |
| Amylase | AMY | U/L | Both | - | + 150 |
| Aspartate transferase | ASTN | IU/L | F | - 30 | + 30 |
| Aspartate transferase | ASTN | IU/L | M | - 30 | + 30 |
| Basophils | BASO | 10 <sup>9</sup> /L | Both | - | + 0.30 |
| Bilirubin conjugated | DBIL | μmol/L | Both | - | + 4.0 |
| Bilirubin total | TBIL | μmol/L | F | - 20.0 | + 10.0 |
| Bilirubin total | TBIL | μmol/L | M | - 20.0 | + 10.0 |
| Bilirubin unconjugated | IBIL | μmol/L | Both | - | - |
| C-reactive protein | CRP | mg/L | Both | - | - |
| CK relative index | CKMBR | % | Both | - | - |
| Calcium | CA | mmol/L | Both | - 0.4 | + 0.4 |
| Carbon dioxide | CO2 | mmol/L | Both | - 8 | + 8 |
| Chloride | CL | mmol/L | Both | - 10 | + 10 |
| Cholesterol | CHOL | mmol/L | Both | - | + 0.7 |
| Creatine kinase | CK | IU/L | F | - | + 400 |
| Creatine kinase | CK | IU/L | M | - | + 400 |
| Creatinine | CREA | μmol/L | Both | - | + 40 |
| Creatinine (DOA urine) | CREDA-U | mmol/L | Both | _ | - |
| Eosinophils | EOS | 10 <sup>9</sup> /L | Both | - | + 0.50 |
| Erythrocyte sedimentation rate | ESR | mm/h | Both | - | - |
| Fibrinogen | FIB-C | g/L | Both | - | - |
| Free T3 | FT3 | pmol/L | Both | - 3.5 | + 3.5 |
| Free T4 | FT4 | pmol/L | Both | - 15.0 | + 15.0 |
| Gamma glutamyl transferase | GGT | IU/L | F | - | + 40 |
| Gamma glutamyl transferase | GGT | IU/L | M | - | + 40 |
| Globulin | GLOB | g/L | Both | - 8 | - |
| Glucose | GLU | mmol/L | Both | - 1.5 | + 2.5 |
| Haematocrit | HCT | L/L | Both | - 0.050 | - |
| Haemoglobin | НВ | g/L | Both | - 20 | - |
| High density lipoprotein | HDL | mmol/L | Both | - 1.50 | + 1.50 |
| International normalised ratio | INRR | ratio | Both | - | - |
| Lactate dehydrogenase | LDH | IU/L | Both | - | + 150 |
| Lymphocytes | LYMP | 10 <sup>9</sup> /L | Both | - 1.50 | + 1.50 |
| Magnesium | MG | mmol/L | Both | - | - |
| Mean cell haemoglobin | МСН | pg | Both | - 2.0 | + 2.0 |
| Mean cell haemoglobin concentration | MCHC | g/L | Both | - 25 | + 25 |
| Mean cell volume | MCV | fL | Both | - 10 | + 10 |

| | | | | Delta | ranges |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable decrease | Acceptable increase |
| Monocytes | MONO | 10 <sup>9</sup> /L | Both | - 0.50 | + 0.50 |
| Neutrophils | NEUT | 10 <sup>9</sup> /L | Both | - 2.00 | + 8.00 |
| Phosphate | PHOS | mmol/L | Both | - 1.00 | + 1.00 |
| Platelets | PLT | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Platelets (citrate tube) | PLTC | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Potassium | K | mmol/L | Both | - 0.8 | + 0.8 |
| Prolactin | PROL | μg/L | Both | | - |
| Prothrombin time | PTT | sec | Both | - 4.0 | + 4.0 |
| Red blood cells | RBC | 10 <sup>12</sup> /L | Both | - 1.0 | - |
| Reticulocyte | RET | % | Both | - | - |
| Reticulocyte count | RETC | 10 <sup>9</sup> /L | Both | - | - |
| Reticulocyte manual count | RETM | 10 <sup>9</sup> /L | Both | - | - |
| Sodium | NA | mmol/L | Both | - 8 | + 8 |
| Thrombin time | TT | sec | Both | - | - |
| Thyroid stimulating hormone | TSH | mIU/L | Both | - 3.00 | + 3.00 |
| Total protein | TP | g/L | Both | - 15 | - |
| Triglycerides | TG | mmol/L | Both | - | + 1.5 |
| Urea | UREA | mmol/L | Both | - 5.0 | + 2.0 |
| Uric acid | UA | μmol/L | Both | - 100 | + 100 |
| Urine pH | UPH | N/A | Both | -4 | + 4 |
| Urine red blood cells | URBC | 10 <sup>6</sup> /L | Both | - | + 10 |
| Urine white blood cells | UWBC | 10 <sup>6</sup> /L | Both | - | + 100 |
| White blood cells | WBC | 10 <sup>9</sup> /L | Both | -2.0 | + 8.0 |

# **Appendix B: Pharmacokinetic Analysis**

#### 1 Calculation Methods

### 1.1 Data Handling Conventions

#### 1.1.1 Actual v Planned Times

Actual sample times will be used for the calculation of pharmacokinetic parameters and for individual concentration-time plots.

Planned sampling times will be used to calculate the concentration-time summary statistics and summary concentration-time plots.

#### 1.1.2 Missing and BQL Concentrations

No missing values will be imputed.

For calculation of all pharmacokinetic parameters and individual profile plots, plasma concentrations below the limit of quantification of the assay (BQL) will be treated as missing (except BQL values observed before the maximum concentration, which will be taken as zero).

BQL values observed post dose will be substituted by one half of the lower limit of quantification for the calculation of concentration summary statistics. Pre dose values will be taken as zero. The number of imputed values will be included in the summary tables.

For urine concentrations reported as BQL it is not possible to impute a value. The amount excreted will be set to zero when concentration is BQL.

#### 1.2 **AUC Calculations**

The AUC will be calculated by a combination of linear and logarithmic methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations.

 $AUC_{(0-\infty)}$  values with <20% of this area extrapolated will be reported.

It is acceptable to include data from profiles with >20% extrapolated as long as at least 80% of the profiles in the study have <20% of the AUC<sub>(0- $\infty$ )</sub> as extrapolated area. In this instance, individual plasma concentration-time profiles for which the extrapolated areas are >20% of AUC<sub>(0- $\infty$ )</sub> will be identified.

It is <u>unacceptable</u> to use  $AUC_{(0-\infty)}$  data if >40% of the AUC has been extrapolated, except in specific situations which should be carefully justified in the study report.

#### 1.3 Lambda-z Calculations

The apparent terminal phase rate-constant ( $\lambda_z$ ) will be estimated by linear regression of logarithmically transformed concentration versus time data. Only those data points which are judged to describe the terminal log-linear decline will be used in the regression.

During the analysis, repeated regressions are carried out using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to  $C_{max}$  are not used. Points with a value of zero for the concentration are excluded. For each regression, an adjusted  $R^2$  is computed. The  $\lambda_z$  using the regression with the largest adjusted  $R^2$  is selected. If the adjusted  $R^2$  does not improve, but is within 0.0001 of the largest adjusted  $R^2$  value, the regression with the larger number of points is used.  $\lambda_z$  must be positive, and calculated from at least three data points.

A minimum number of three data points will be used in calculating  $\lambda_z$ .

For non-compartmental analysis uniform weighting will be applied.

If non-linear regression (i.e. compartmental) analysis is used then weighting by y<sup>-1</sup> or y<sup>-2</sup> should be investigated.

Justification for rule: The log transformation of the data in calculation of  $\lambda_z$  sufficiently deals with the heterogeneous variability of the concentration data and no further weighting is necessary.

#### 1.4 Observed v Predicted Values

For parameters dependent on  $\lambda_z$ , the 'predicted' rather than the 'observed' parameters will be calculated.

The 'predicted' parameters are calculated using  $\hat{C}_{\iota}$  (the predicted value of the concentration at time tn); whilst the 'observed' parameters use the last observed concentration.

# 2 General Considerations for Data Analysis

#### 2.1 Derived and transformed data

A list of those parameters that will be log transformed will be given in the SAP.

In general, concentration and concentration-related quantities, rate constants and half-lives (e.g.  $C_{max}$ , AUC,  $t_{1/2}$ , CL/F,  $V_z$ /F and MRT) will be analysed after logarithmic transformation. Logarithmic transformations will use natural logarithms (log<sub>e</sub>).

If t<sub>max</sub> is subjected to a statistical analysis, it will not be transformed and will be analysed using non-parametric methods (Cartwright et al.(1991)).

# 2.2 Summary data

Means at any time will only be calculated if at least 2/3 of the individual data are measured and are above the lower limit of quantification (LLOQ).

# 3 Parameter Definitions

# 3.1 Plasma Parameters

## 3.1.1 Single Dose

Emodepside parameters to be calculated on Day 0.

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Concentrations an | | | | | | | |
| C <sub>max</sub> | Maximum (peak) plasma concentration | The maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | ng/mL | Y | Cmax | CMAX | C <sub>max</sub> |
| C <sub>max</sub> /Dose | Dose-normalised AUC to infinity | The dose-normalised C <sub>max</sub> will be calculated as C <sub>max</sub> /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | C <sub>max</sub> /D |
| C <sub>max,norm</sub> | Observed maximum plasma concentration corrected by dose and body weight | The C <sub>max</sub> normalised by dose and body weight will be calculated as C <sub>max</sub> /(Dose administered*body weight) | (ng/mL)/(mg*kg) | Y | <u>-</u> | CMAXWD | Cmax,norm |
| t <sub>max</sub> | Time to reach maximum (peak) plasma concentration | The first time of maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | h | N | Tmax | TMAX | t <sub>max</sub> |
| Areas under the ci | urve | | | | | | |
| AUC <sub>12</sub> * | Area under the plasma concentration-time curve from time zero to time 12 h | The area under the concentration-time curve from zero time (pre-dose) to time 12 h will be calculated using the (specified) trapezoidal method. If $\lambda_z$ is not estimable, a partial AUC is not | h*ng/mĽ | Y | User specified area | AUCINT | AUC <sub>12</sub> |
| AUC <sub>12</sub> /Dose * | Dose-normalised AUC from time zero to 12 h | calculated (when t <sub>last</sub> <t). 12h="" as="" auc="" auc<sub="" be="" calculated="" dose-normalised="" from="" the="" time="" to="" will="" zero="">12/Dose Administered</t).> | (h*ng/mL)/mg | Y | - | AUCINTD | AUC <sub>12</sub> /D |
| AUC12,norm* | Area under the concentration-time curve from time zero to 12h corrected by dose and body | The AUC from time zero to 12h normalised by dose and body weight will be calculated as AUC12/(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | - | AUCINTWD | AUC <sub>12,norm</sub> |

| Text Symbol | Definition<br>weight | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| AUC <sub>24</sub> ** | Area under the plasma concentration-time curve from time zero to time 24 h | The area under the concentration-time curve from zero time (pre-dose) to time 24 h will be calculated using the (specified) trapezoidal method. | h*ng/mL | Y | User specified area | AUCINT | AUC <sub>24</sub> |
| | | If $\lambda_z$ is not estimable, a partial AUC is not calculated (when $t_{last} < t$ ). | | | | | |
| AUC <sub>24</sub> /Dose ** | Dose-normalised AUC from time zero to 24 h | The dose-normalised AUC from time zero to 24h will be calculated as AUC24/Dose Administered | (h*ng/mL)/mg | Y | - | AUCINTD | AUC <sub>24</sub> /D |
| AUC24,norm ** | Area under the concentration-time curve from time zero to 24h corrected by dose and body weight | The AUC from time zero to 24h normalised by dose and body weight will be calculated as AUC24/(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | - | AUCINTWD | AUC <sub>24,norm</sub> |
| Clearance, volume | of distribution and mean resid | lence time | | | | · · · · · · · | |
| V <sub>z</sub> /F | Apparent volume of distribution during terminal phase after non-intravenous administration | Apparent volume of distribution will be calculated using the following formula: $V_z/F = \frac{Dose}{\lambda_z \bullet AUC_{\infty}}$ | L | Y | Vz_pred (actually derives Vz_F_pred for oral dose) | VZFP | V₂/F |
| MRT <sub>last</sub> | Mean Residence Time | The mean residence time will be calculated using: $MRT = \frac{AUMC}{AUC_{\infty}}$ | h | Y | MRTLST_pred | MRTEVLST | MRT <sub>last</sub> |

<sup>\*</sup> Calculated only for Cohort 3

<sup>\*\*</sup>Calculated only for Cohorts 1 and 2

# 3.1.2 Multiple Dose

Emodepside parameters to be calculated on Day 9.

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| | ring and after multiple dosing | | | | | | |
| C <sub>trough</sub> | Trough plasma concentration | Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration]) obtained directly from the concentration-time data. | ng/mL | Y | - | CTROUGH | C <sub>trough</sub> |
| Concentrations and | d times (after final dose) | | | | | | |
| C <sub>max,ss</sub> | Maximum (peak) plasma concentration at steady state | The maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | ng/mL | Y | Cmax | CMAX | $C_{max,ss}$ |
| C <sub>max,ss</sub> /Dose | Dose-normalised C <sub>max</sub> at steady state | The dose-normalised C <sub>max</sub> will be calculated as C <sub>max</sub> /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | C <sub>max.ss</sub> /D |
| C <sub>max,ss,norm</sub> | Observed maximum plasma concentration corrected by dose and body weight at steady state | The C <sub>max</sub> normalised by dose and body weight will be calculated as C <sub>max</sub> /(Dose administered*body weight) | (ng/mL)/(mg*kg) | Y | • | CMAXWD | Cmax,ss,norm |
| t <sub>max</sub> | Time to reach maximum (peak) plasma concentration | The first time of maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | h | N | Tmax | TMAX | t <sub>max</sub> |
| Half-life (after fina | ıl dose) | | | | | | |
| $\lambda_{z}$ | Terminal rate constant | The apparent terminal phase rate-constant $(\lambda_2)$ will be estimated by linear regression of logarithmically transformed concentration versus time data. | 1/h | Y | Lambda_z | LAMZ | λ <sub>z</sub> |
| t <sub>1/2</sub> | Terminal half-life | The terminal half-life calculated from the terminal slope of the log concentration-time curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | LAMZHL | t <sub>1/2</sub> |
| t <sub>½,dom</sub> | Dominant half-life | The dominant half-life calculated from the terminal slope of the log concentration-time (0-24h) curve, as follows: | h | Y | HL_Lambda_z | LAMZHLD | t1/2,0-24 |

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| | | $t_{1/2}, dom = \frac{\log_{\sigma} 2}{\lambda_{z}}$ | | , | | | |
| | rve (after final dose) | | , | · | | | |
| AUC <sub>last</sub> | Area under the plasma concentration-time curve from time zero to time of last measurable concentration | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration will be calculated using the (specified) trapezoidal method. | h*ng/mL | Y | AUClast | AUCLST | AUC <sub>last</sub> |
| AUC <sub>last</sub> /Dose | Dose-normalised AUC from time zero to last measurable concentration | The dose-normalised AUC from time zero to last measurable concentration will be calculated as AUClast/Dose Administered | (h*ng/mL)/mg | Y | • | AUCLSTD | AUC <sub>last</sub> /D |
| AUC <sub>last,norm</sub> | Area under the concentration-time curve from time zero to time of last measurable concentration corrected by dose and body weight | The AUC from time zero to last measurable concentration normalised by dose and body weight will be calculated as AUClast/(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | <u>-</u> | AUCLSTWD | AUC <sub>last,norm</sub> |
| AUC <sub>12</sub> * | Area under the plasma concentration-time curve from time zero to time 12 h | The area under the concentration-time curve from zero time (pre-dose) to time 12 h will be calculated using the (specified) trapezoidal method. If λ <sub>z</sub> is not estimable, a partial AUC is not calculated (when t <sub>last</sub> <t).< td=""><td>h*ng/mL</td><td>Y</td><td>User specified area</td><td>AUCINT</td><td>AUC<sub>12</sub></td></t).<> | h*ng/mL | Y | User specified area | AUCINT | AUC <sub>12</sub> |
| AUC <sub>12</sub> /Dose * | Dose-normalised AUC from time zero to 12 h | The dose-normalised AUC from time zero to 12h will be calculated as AUC <sub>12</sub> /Dose Administered | (h*ng/mL)/mg | Y | - | AUCINTD | AUC <sub>12</sub> /D |
| AUC12,norm * | Area under the concentration-time curve from time zero to 12h corrected by dose and body weight | The AUC from time zero to 12h normalised by dose and body weight will be calculated as AUC12/(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | - | AUCINTWD | AUC <sub>12,norm</sub> |

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| AUC <sub>24</sub> ** | Area under the plasma concentration-time curve from time zero to time 24 h | The area under the concentration-time curve from zero time (pre-dose) to time 24 h will be calculated using the (specified) trapezoidal method. If $\lambda_z$ is not estimable, a partial AUC is not calculated (when $t_{last} < t$ ). | h*ng/mL | Y | User specified area | AUCINT | AUC <sub>24</sub> |
| AUC <sub>24</sub> /Dose ** | Dose-normalised AUC from time zero to 24 h | The dose-normalised AUC from time zero to 24h will be calculated as AUC24/Dose Administered | (h*ng/mL)/mg | Y | - | AUCINTD | AUC <sub>24</sub> /D |
| AUC24,norm ** | Area under the concentration-time curve from time zero to 24h corrected by dose and body weight | The AUC from time zero to 24h normalised by dose and body weight will be calculated as AUC24/(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | | AUCINTWD | AUC <sub>24,norm</sub> |

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| AUC∞ | Area under the plasma concentration-time curve from time zero to infinity | The area under the concentration-time curve will be calculated using the (specified) trapezoidal method for the interval 0 to $t_{last}$ (time $t_{last}$ is the time at which the last non-zero level was recorded), plus the area under the exponential curve from $t_{last}$ to infinity, calculated as follows: $AUC_{t-\infty} = \frac{\hat{C}_t}{\lambda_z} \text{where } \hat{C}_t \text{ is the predicted value of the concentration at } t_{last}.$ | h*ng/mL | Y | AUCINF_pred | AUCIFP | AUC <sub>inf</sub> |
| AUC <sub>&amp;</sub> /Dose | Dose-normalised AUC from time zero to infinity | The dose-normalised AUC from time zero to infinity will be calculated as AUC <sub>∞</sub> /Dose Administered | (h*ng/mL)/mg | Y | - | AUCIFPD | AUC <sub>∞</sub> /D |
| $\mathrm{AUC}_{\infty,\mathrm{norm}}$ | Area under the concentration-time curve from time zero to infinity corrected by dose and body weight | The AUC from time zero to infinity normalised by dose and body weight will be calculated as AUC <sub>\omega</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | - | AUCIFPWD | AUC <sub>∞,norm</sub> |
| %AUC <sub>extrap</sub> | Percentage of $AUC_{\infty}$ extrapolated from from $t_{last}$ to infinity | $\%AUC_{extrap} = \frac{100 \times AUC_{t-x}}{AUC_{x}}$ | % | N | AUC_%EXTRAP_pr<br>ed | AUCPEP | %AUC <sub>extrap</sub> |
| learance, volume ( | of distribution and mean resider | nce time (after final dose) | | | | - | |
| CL <sub>SS</sub> /F | Apparent total clearance from plasma after oral administration | Apparent total clearance from plasma will be calculated using the following formula: $CL_{SS} / F = \frac{Dose}{AUC_{r}}$ | L∕h | Y | Clss_pred (actually derives Clss_F_pred for oral dose) | CLFTAU | CL <sub>SS</sub> /F |
| V <sub>2</sub> /F | Apparent volume of distribution after non-intravenous administration calculated at steady state | Apparent volume of distribution calculated at steady state will be calculated using the following formula: $V_z / F = \frac{Dose}{\lambda_z \bullet AUC_\tau}$ | L | Y | Vz_pred (actually derives Vz_F_pred for oral dose) | VZFTAU | V <sub>z</sub> /F |

Sponsor code: DNDI-EMO-02

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| MRT∞ | Mean Residence Time extrapolated to infinity | The mean residence time will be calculated using: | h | Y | MRTINF_pred | MRTEVIFP | MRT <sub>∞</sub> |
| Accumulation and t | ime invariance ratios | $MRT = \frac{AUMC}{AUC_{\infty}}$ | | | | | |
| R <sub>ac(</sub> AUC) | Accumulation ratio for AUC | Accumulation ratio will be calculated from AUC, at steady state and AUC, after single dose | - | N | - | ARAUC | R <sub>ac(</sub> AUC) |
| R <sub>ac(</sub> C <sub>max)</sub> | Accumulation ratio for C <sub>max</sub> | Accumulation ratio will be calculated from $C_{max}$ at steady state and $C_{max}$ after single dose | - | N | - | ARCMAX | R <sub>ac(</sub> C <sub>max)</sub> |

<sup>\*</sup> Calculated only for Cohort 3

<sup>\*\*</sup>Calculated only for Cohorts 1 and 2

Sponsor code: DNDI-EMO-02

# **Appendix C: Sample Page Layout**

| DNDi: DNDI-EMO-02 Cohorts | Page x of y | |
|---|---|---|
| Population: [Pop] | | |
| | Table [number] [title] | |
| | Column headers | - |
| | Main body of output | _ |
| | Source: Listing [16.2.xx] | _ |
| Footnotes about the table or l | isting text go here. | |
| Program: [Prog Name] Produced By:[Username] | [Date] | HMR: 16-021 Cohorts 1 and 2 |
| i roduced by.[Osemaine] | | |

Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"

<sup>\*</sup>y = last page of individual output